CLINICAL TRIAL: NCT03408067
Title: "Evaluation of the Efficacy of Two Nutritional Risk Screening Tests, Nutritional Risk Screening 2002 (NRS 2002) and Subjective Global Assessment (SGA), to Identifying Malnourished or at Risk of Malnutrition Hospital Patients"
Brief Title: Evaluation of the Efficacy of Nutritional Risk Screening Tests, NRS 2002 and SGA, to Identifying Malnourished Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Fabrizio Pasanisi, MD, Federico II University
Other Study IDs: 164/16
Record Dates: First submitted 2017-12-19; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In several hospital clinical trials, the nutritional intervention has been proven to be effective in preventing and/or reducing malnutrition. Therefore, a procedure to identify the risk of malnutrition or malnourishment in hospitalized patients is necessary to guarantee an adequate and timely nutritional treatment.

Aims: to compare two validated nutritional screening tools: NRS 2002 and SGA. These are used to identify the risk of malnutrition or malnourishment in hospitalized patients.

Patients and Methods: The study is currently carried out at the Federico II University Hospital of Naples, Italy. The in patients admitted in the Clinical Wards since September 2016 are being evaluated. The two screening test results and the assessment of the patients' parameters are collected within 72 hours following admission. Age, sex, height, weight, Body Mass Index (BMI), calf circumference and dominant hand of the participants are being noted. Venous blood samples are collected for routine biochemistry and inflammatory parameters ; all measurements are determined by routine laboratory methods at the Department of Laboratory Medicine of the University Hospital Federico II, Naples.

DETAILED DESCRIPTION:
In several hospital clinical trials, the nutritional intervention has been proven to be effective in preventing and/or reducing malnutrition. Therefore, a procedure to identify the risk of malnutrition or malnourishment in hospitalized patients is necessary to guarantee an adequate and timely nutritional treatment. It is mandatory for clinics and health services to perform the screening test for the evaluation of the nutritional status and need in hospitalized patient.

Aims: The first aim of this study is to compare two validated nutritional screening tools: Nutritional Risk Screening 2002 (NRS 2002) and Subjective Global Assessment (SGA). These are used to identify the risk of malnutrition or malnourishment in hospitalized patients. The second aim is to evaluate possible correlations between the tests score and body composition parameters (phase angle of the Bioelectrical Impedance Analysis, BIA), handgrip strength and biochemical parameters.

Patients and Methods: The study is currently carried out at the Federico II University Hospital of Naples, Italy. The inpatients admitted in the Clinical Wards coming from the Emergency Room of the Hospital since September 2016 are being evaluated. The two screening test results and the assessment of the patients' parameters are collected within 72 hours following admission. The SGA and NRS 2002 are administered separately. Age, sex, height, weight, Body Mass Index (BMI), calf circumference and dominant hand of the participants are being noted. Venous blood samples are collected for routine biochemistry and inflammatory parameters (C-reactive protein, fibrinogen) early in the morning in the fasting state; all measurements are determined by routine laboratory methods at the Department of Laboratory Medicine of the University Hospital Federico II, Naples.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years.

Exclusion Criteria:

* Inpatients of the intensive care unit after admission from Emergency Room;
* Pregnancy and breastfeeding.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hospital Wards inpatients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
malnutrition scored with NRS 2002 questionnaire | 5 minutes
  scoring scale (units 0-3) : 0 = nourished patient; 1 = mild malnutrition, 2 = moderate malnutrition, 3 = severe malnutrition
malnutrition scored with SGA questionnaire | 5 minutes
  scoring scale (units a-c) : a = nourished patient; b = mildly malnourished; c = severely malnourished

CONTACTS AND LOCATIONS:
Locations (1):
- Fabrizio Pasanisi, Napoli, Italy

IPD SHARING:
Plan to Share IPD: Undecided